CLINICAL TRIAL: NCT02057965
Title: Autologous Bone Marrow Derived Mesenchymal Stromal Cell Therapy in Combination With Everolimus to Preserve Renal Structure and Function in Renal Recipients
Brief Title: Mesenchymal Stromal Cell Therapy in Renal Recipients
Acronym: MSCs
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, M.E. J. Reinders, MD/PhD, Leiden University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL43712.000.13; 2013-000819-25 (EudraCT Number)
Record Dates: First submitted 2014-02-05; First posted 2014-02-07 (Estimated); Last update posted 2020-09-17 (Actual); Status verified 2020-09

CONDITIONS: Renal Transplant Rejection; Fibrosis
Keywords: Mesenchymal Stromal Cells; Allograft rejection; Fibrosis
MeSH Terms: conditions — Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mesenchymal Stromal Cells + Everolimus (Active Comparator): Intervention: two doses of autologous bone marrow (BM) derived Mesenchymal Stromal Cells IV, 7 days apart, 6 and 7 weeks after transplantation in combination with Certican® (1.5mg/day). Doses of MSCs will be 1-2x10^6 million MSCs per/kg body weight.
  At the time of the second MSC infusion tacrolimus will be withdrawn in 2 weeks (after 1 week dose of tacrolimus wil be halved, after 2 weeks stopped)
  Interventions: Drug: Mesenchymal Stromal Cells
- Everolimus + Tacrolimus (No Intervention): Patients in the control group will receive Certican® (1.5 mg b.i.d.) and standard dose tacrolimus (through levels 6-8 ng/ml after 6 weeks).

INTERVENTIONS:
Drug: Mesenchymal Stromal Cells — Two doses of autologous bone marrow (BM) derived MSCs IV, 7 days apart, 6 and 7 weeks after transplantation. Doses of MSCs will be 1-2x10^6 million MSCs per/kg body weight
  Other Names: Bone marrow derived mesenchymal stromal cells
  Arms: Mesenchymal Stromal Cells + Everolimus

SUMMARY:
This study will test the hypothesis that MSCs in combination with Everolimus facilitate Tacrolimus withdrawal, reduce fibrosis and decrease the incidence of opportunistic infections compared to standard tacrolimus dose.

DETAILED DESCRIPTION:
Kidney transplantation has improved survival and quality of life for patients with end-stage renal disease. Despite excellent short-term results, long-term survival of transplanted kidneys has not improved accordingly in the last decades. Calcineurin inhibitors (CNI) have been the cornerstone of immunosuppressive therapy for many years, due to their efficacy in preventing acute rejection. However, CNI have nephrotoxic side effects that can directly contribute to renal dysfunction and compromise long-term outcomes. Consequently there is a strong interest in immunosuppressive (IS) regimens that maintain efficacy for the prevention of acute rejection, whilst reducing nephrotoxicity.

In this perspective the combination of mesenchymal stromal cells (MSCs) with a mTor inhibitor (Everolimus (Certican®)) might be an optimal strategy to facilitate CNI (tacrolimus) withdrawal. MSCs have IS properties and roles in tissue repair and everolimus is a proliferation signal inhibitor with potent immunosuppressant effects. In experimental studies the combination of mTor inhibitor and MSCs was shown to attenuate alloimmune responses and to promote allograft tolerance.

In total 70 de novo renal recipients, 18-75 years of ages will be recruited from the transplant clinics of the LUMC. Thirty five of these patients will be included in the Certican/ and MSC group and 35 patients in the Certican/ standard dose tacrolimus group. Patients of the MSC treated groups will receive two doses of autologous BM derived MSCs IV, 7 days apart, 6 and 7 weeks after transplantation in combination with Certican® (1.5 mg b.i.d.). At the time of the second MSC infusion tacrolimus will be withdrawn in 2 weeks (after 1 week dose of tacrolimus will be halved, after 2 weeks stopped). Patients in the control group will receive Certican® (1.5 mg b.i.d.) and standard dose tacrolimus (through levels 6-8 ng/ml after 6 weeks).

Primary goal is evaluate whether concentration-controlled Certican® with MSCs compared to Certican® with standard tacrolimus in renal transplant recipients reduces fibrosis by quantitative Sirius Red scoring.

ELIGIBILITY:
Inclusion Criteria:

* Subject is willing to participate in the study, must be able to give informed consent and the consent must be obtained prior to any study procedure.
* Recipients of a first kidney graft from a deceased, living-unrelated or non-HLA identical living related donor > 50 years of age.
* Panel Reactive Antibodies (PRA) ≤ 10%.
* Patients must be able to adhere to the study visit schedule and protocol requirements.
* If female and of child-bearing age, subject must be non-pregnant, non-breastfeeding, and use adequate contraception.

Exclusion Criteria:

* Double organ transplant recipient.
* Biopsy proven acute rejection (according to the Banff criteria) in the first 6 weeks after transplantation.
* Patients with evidence of active infection or abscesses (with the exception of an uncomplicated urinary tract infection) before MSC infusion.
* Patients suffering from hepatic failure.
* Patients suffering from an active autoimmune disease.
* Patients who have had a previous BM transplant.
* A psychiatric, addictive or any disorder that compromises ability to give truly informed consent for participation in this study.
* Use of any investigational drug after transplantation.
* Documented HIV infection, active hepatitis B, hepatitis C or TB according to current transplantation inclusion criteria.
* Subjects who currently an active opportunistic infection at the time of MSC infusion (e.g., herpes zoster [shingles], cytomegalovirus (CMV), Pneumocystis carinii (PCP), aspergillosis, histoplasmosis, or mycobacteria other than TB, BK) after transplantation.
* Malignancy (including lymphoproliferative disease) within the past 2-5 years (except for squamous or basal cell carcinoma of the skin that has been treated with no evidence of recurrence) according to current transplantation inclusion criteria.
* Known recent substance abuse (drug or alcohol).
* Contraindications to undergo a BM biopsy.
* Patients who are recipients of ABO incompatible transplants.
* Cold ischemia time >30 hrs.
* Patients with severe total hypercholesterolemia (>7.5 mmol/L) or total hypertriglyceridemia (>5.6 mmol/L) (patients on lipid lowering treatment with controlled hyperlipidemia are acceptable).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2014-03; Primary Completion 2020-01 (Actual); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Fibrosis by quantitative Sirius Red scoring of MSC treated and untreated groups | at 6 months compared to 4 weeks post transplant

SECONDARY OUTCOMES:
Renal function and proteinuria | 6 months
Number of participants with CMV and BK infection an other opportunistic infections between groups | 6 months
Number of participants with adverse events | 6 months
composite end point efficacy failure (biopsy proven acute rejection, graft loss or death) | 6 months
Presence of donor specific antibodies and immunologic monitoring | 6 months
Progression of subclinical cardiovascular disease in the different treatment groups bij assessing echocardiographic parameters | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Marlies EJ Reinders, MD/PhD, Principal Investigator — Leiden University Medical Center
Locations (1):
- Leiden University Medical Center, Leiden, Netherlands

REFERENCES:
- [Result] Reinders ME, de Fijter JW, Roelofs H, Bajema IM, de Vries DK, Schaapherder AF, Claas FH, van Miert PP, Roelen DL, van Kooten C, Fibbe WE, Rabelink TJ. Autologous bone marrow-derived mesenchymal stromal cells for the treatment of allograft rejection after renal transplantation: results of a phase I study. Stem Cells Transl Med. 2013 Feb;2(2):107-11. doi: 10.5966/sctm.2012-0114. Epub 2013 Jan 24. PMID 23349326
- [Derived] Hendriks SH, Heidt S, Schulz AR, de Fijter JW, Reinders MEJ, Koning F, van Kooten C. Peripheral Blood Immune Cell Composition After Autologous MSC Infusion in Kidney Transplantation Recipients. Transpl Int. 2023 Jun 23;36:11329. doi: 10.3389/ti.2023.11329. eCollection 2023. PMID 37426430
- [Derived] Reinders ME, Bank JR, Dreyer GJ, Roelofs H, Heidt S, Roelen DL, Al Huurman V, Lindeman J, van Kooten C, Claas FH, Fibbe WE, Rabelink TJ, de Fijter JW. Autologous bone marrow derived mesenchymal stromal cell therapy in combination with everolimus to preserve renal structure and function in renal transplant recipients. J Transl Med. 2014 Dec 10;12:331. doi: 10.1186/s12967-014-0331-x. PMID 25491391